CLINICAL TRIAL: NCT03092414
Title: CMV Criteria in the Detection of Gastric Diseases Using Linked Color Imaging
Brief Title: Linked Color Imaging Based CMV Diagnosis for Gastric Mucosal Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 307-LCI-004
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Gastric Disease
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients with indications for gastroduodenoscopy will be evaluated with WLE and then LCI.
  Interventions: Procedure: WLE and then LCI
- Group B (Experimental): Patients with indications for gastroduodenoscopy will be evaluated with LCI and then WLE.
  Interventions: Procedure: LCI and then WLE

INTERVENTIONS:
Procedure: WLE and then LCI — The gastric mucosa was evaluated with WLE and then LCI by two different endoscopists.
  Arms: Group A
Procedure: LCI and then WLE — The gastric mucosa was evaluated with LCI and then WLE by two different endoscopists.
  Arms: Group B

SUMMARY:
The newly developed linked color imaging (LCI) system (FUJIFILM Co.) creates clear and bright endoscopic images by using short-wavelength narrow-band laser light combined with white laser light on the basis of BLI technology. This system can obtain bright endoscopic images even at a distant view because LCI has more intense white light than the short-wavelength narrow-band laser light. Short-wavelength narrow-band laser light enhances the vessels on the mucosal surface and the patterns of the mucosa. Therefore, LCI may facilitate the detection of gastric mucosal lesions. Further studies are needed to confirm the clinical utility of LCI.

DETAILED DESCRIPTION:
LCI enhances differences in hue, in the red region of the spectrum, through digital processing. This makes red areas appear redder and white areas appear whiter. Thus, it is easier to recognize a slight difference in color of the mucosa. Based on previous experience, a new LCI based endoscopic diagnosis criteria called CMV (color- microstructure-vessel) criteria has been proposed, which could be used for judging the gastric mucosal lesions. LCI has the advantage of detecting color changes of the mucosa, and this could provide very valuable and useful evidence for making endoscopic diagnosis. In this study, a blinded random controlled clinical trial is designed to further validate the diagnostic value of LCI based CMV criteria for gastric diseases.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old patients
* Who agree to participate in the study
* Patients with the indications for gastroduodenoscopy

Exclusion Criteria:

* Patients, who were receiving nonsteroidal anti-inflammatory drugs, pump inhibitors (PPI) or antibiotics in the last 3 weeks.
* Severe uncontrolled coagulopathy
* Prior history of gastric surgery.
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 4 months
  Diagnostic accuracy of LCI for gastric diseases was calculated by comparing the LCI endoscopic diagnosis with pathological diagnosis.

SECONDARY OUTCOMES:
Numbers of lesions in the stomach | 4 months
  The numbers of lesion detected under WLE and LCI will be recorded and compared.
Endoscopic examination duration | 4 months
  The time spent on the endoscopic examination using WLE and LCI will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, M.D., Ph.D., Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital to Academy of Military Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun X, Dong T, Bi Y, Min M, Shen W, Xu Y, Liu Y. Linked color imaging application for improving the endoscopic diagnosis accuracy: a pilot study. Sci Rep. 2016 Sep 19;6:33473. doi: 10.1038/srep33473. PMID 27641243
- [Background] Dohi O, Yagi N, Onozawa Y, Kimura-Tsuchiya R, Majima A, Kitaichi T, Horii Y, Suzuki K, Tomie A, Okayama T, Yoshida N, Kamada K, Katada K, Uchiyama K, Ishikawa T, Takagi T, Handa O, Konishi H, Naito Y, Itoh Y. Linked color imaging improves endoscopic diagnosis of active Helicobacter pylori infection. Endosc Int Open. 2016 Jul;4(7):E800-5. doi: 10.1055/s-0042-109049. PMID 27556101
- [Background] Ono S, Abiko S, Kato M. Linked color imaging enhances gastric cancer in gastric intestinal metaplasia. Dig Endosc. 2017 Mar;29(2):230-231. doi: 10.1111/den.12757. Epub 2016 Nov 21. No abstract available. PMID 27770584
- [Derived] Min M, Dong TH, Liu Y, Bi YL, Ma CY. Novel endoscopic findings as visualized by non-magnification endoscopy with linked color imaging are indicative of gastric intestinal metaplasia. Chin Med J (Engl). 2019 Apr 5;132(7):782-788. doi: 10.1097/CM9.0000000000000172. PMID 30896610